CLINICAL TRIAL: NCT07334691
Title: "TARGET 2.0 Study": Safety and Performance of the Cardiovalve Tricuspid Valve Replacement System in the Treatment of Subjects With Tricuspid Regurgitation- Investigation
Brief Title: "TARGET 2.0 Study": Safety and Performance of the Cardiovalve TR Replacement System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiovalve Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-25-01
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiovalve TR valve replacement System (Experimental): The Cardiovalve system includes a valve and delivery system, designed for replacement of the tricuspid valve through a transcatheter.
  Interventions: Device: Cardiovalve TR valve replacement System

INTERVENTIONS:
Device: Cardiovalve TR valve replacement System — Cardiovalve Tricuspid Valve Replacement system

SUMMARY:
This investigation is a continuation for "TARGET" investigation and its purpose is to further demonstrate the efficiency and safety of the Cardiovalve system in the treatment of subjects with tricuspid regurgitation. The same subject population will be included, while applying the clinical and scientific knowledge accumulated in the TARGET investigation. This investigation will support the submission for obtaining marketing approval.

DETAILED DESCRIPTION:
"TARGET 2.0": Safety and Performance of the Cardiovalve Tricuspid valve replacement system in the treatment of subjects with tricuspid regurgitation- investigation: Cardiovalve Tricuspid Valve Replacement system (hereinafter referred to as Cardiovalve TR system) The system has not been granted CE mark at this time The Cardiovalve implant consists of three bovine pericardium tissue leaflets, self-expanding dual nitinol frame, and fabric. A total of 24 anchoring points affix the device to the native tricuspid annulus.

The Delivery System is intended to deliver the valve in the crimped position via the transfemoral venous approach. It comprises of a catheter assembly and handles. The handles knobs facilitate valve alignment and positioning in the native valve, and control the capsule expansion and release of the Cardiovalve implant.

The Cardiovalve TR Valve Replacement System is intended for reduction of tricuspid regurgitation (TR) in patients with symptomatic severe or greater secondary tricuspid regurgitation despite being treated with medical therapy for whom tricuspid valve replacement is deemed appropriate by a Heart Team. The system percutaneously delivers the Implant to the tricuspid valve via femoral vein access This investigation is a continuation for "TARGET" investigation and its purpose is to further demonstrate the efficiency and safety of the Cardiovalve system in the treatment of subjects with tricuspid regurgitation. The same subject population will be included, while applying the clinical and scientific knowledge accumulated in the TARGET investigation. This investigation will support the submission for obtaining marketing approval.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 and <85 years
2. Severe tricuspid regurgitation (TR) ≥3+ based upon echocardiography, as assessed by independent core laboratory using a 5-grade classification (mild (1), moderate (2), severe (3), massive (4), torrential (5)). Trace and no TR is considered 0)29
3. Symptomatic, NYHA Class II-IV
4. Left ventricular ejection fraction (LVEF) ≥ 30%
5. Subject adequately treated based upon medical standards
6. Subjects are at high risk for open heart surgery
7. Subject provided written, informed consent before investigation enrollment
8. Subject approved by the Subject Screening Committee

   Anatomical Inclusion Criteria (measured by CT)
9. Right femoral vein diameter > 9mm
10. Tricuspid valve diameter < 55 mm
11. RV length > 45 mm

Exclusion Criteria:

Subjects will be excluded from the investigation if fulfill any of the following criteria:

1. Cardiac anatomy deemed not suitable for the Cardiovalve TR system as evaluated (by CT)
2. Venous peripheral anatomy or any spinal anatomy that is unsuitable for Cardiovalve TR implant delivery (by CT)
3. Primary tricuspid disease that may interfere with Cardiovalve implantation
4. Severe right ventricular failure (by Echo core lab adjudication)
5. Significant coronary artery disease requiring percutaneous or surgical intervention
6. Severe systolic pulmonary arterial pressure, pASP > 2/3 systemic BP with PVR > 5 Wood units after vasodilator challenge
7. Presence of any known life threatening non-cardiac disease that will limit the subject's life expectancy to less than one year
8. Cerebrovascular event (stroke, TIA) within the past 3 months
9. Active endocarditis or history of mitral/tricuspid endocarditis within 3 months or infection requiring antibiotic within 2 weeks before index procedure
10. Subject has significant other sided valvular heart disease which requires treatment (e.g. mitral regurgitation or stenosis, or aortic regurgitation or stenosis)
11. Documented primary coagulopathy or platelet disorder, including thrombocytopenia (absolute platelet count <90k)
12. Documented evidence of significant renal dysfunction (eGFR<30 ml/min/1.73m2) or any form of dialysis at time of screening within 30 days
13. Untreatable hypersensitivity or contraindication to any of the following: all antiplatelets, all anticoagulants, nitinol alloys (nickel and titanium), bovine tissue, glutaraldehyde, contrast media, or Polyethylene Glycol (PEG)
14. Subjects unsuitable for implantation due to thrombosis of the lower venous system or presence of a vena cava filter
15. Evidence of an acute myocardial infarction (AMI) ≤ 1 month (30 days)
16. Liver cirrhosis > Child-Pugh Class A
17. Psychiatric or behavioral disease including known alcohol or drug abuser that is likely to impair compliance with protocol
18. Pregnant, lactating or planning pregnancy within next 12 months
19. Requirement for antibiotic treatment within the last 48 hours
20. Surgical or interventional procedure planned within 30 days prior to index procedure
21. Refractory heart failure requiring advanced intervention (i.e. left ventricular assist device, transplantation) or UNOS Status 1 heart transplant or prior orthotropic heart transplantation.
22. Prior Tricuspid valve surgery or transcatheter tricuspid valve procedure that may interfere with the Cardiovalve device. Valve in a valve procedure is excluded.
23. Modified Rankin Scale > 4 disability
24. Implant or revision of any rhythm management device (CRT or CRT-D) or implantable cardioverter-defibrillator within 30 days prior to index procedure
25. Acutely decompensated heart failure (i.e. hemodynamically unstable or requiring IV inotrope) at the time of screening
26. Severe COPD or continuous use of home oxygen
27. Hgb < 9 g/dL at screening
28. The subject has contraindication against a transesophageal echo (TEE) during the procedure that cannot be replaced by other imaging.
29. Currently participating in an investigational drug or another device investigation which has not reached its primary endpoint
30. Subjects with >2 leads or with any lead that may interfere with Cardiovalve procedure or device

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2033-09 (Estimated)

PRIMARY OUTCOMES:
Freedom from device or procedure-related adverse events | 30 days
  Freedom from device or procedure-related adverse events
Reduction in TR grade | 30 days
  Reduction in TR in comparison to baseline

SECONDARY OUTCOMES:
Six minute walk test | 30 days, 6 months, 12 months, annual for five years
  Change in Six minute walk distance from Baseline
KCCQ | 30 days, 6 months, 12 months, annual for five years
  Change in health status from Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Georg Nickenig, Principal Investigator — Bonn Clinic
Locations (2):
- Germany (2):
  - Uniklinik Bonn -, Bonn
  - Bonn Clinic, Bonn

IPD SHARING:
Plan to Share IPD: No
No plan